CLINICAL TRIAL: NCT03928457
Title: Impact of Chronic Exposure to Radiofrequency Electromagnetic Fields on Neurophysiological Development in the Preterm Neonate
Acronym: NeuroPrem-RF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PI2018_843_0033
Record Dates: First submitted 2019-04-16; First posted 2019-04-26 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Preterm Infant; Exposure to Radiofrequency
Keywords: preterm neonate; radiofrequency exposure; neurophysiological functions
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- preterm neonate (Experimental)
  Interventions: Other: Parental questionnaire; Other: Daily continuous recording of radiofrequency exposure levels; Other: Follow-up of daily infants environmental and clinical parameters; Other: Nocturnal polysomnography; Diagnostic Test: cerebral hemodynamics; Diagnostic Test: activity of the autonomic nervous system

INTERVENTIONS:
Other: Parental questionnaire — Parental questionnaire on pregnancy history and environmental exposure
Other: Daily continuous recording of radiofrequency exposure levels — Daily continuous recording of radiofrequency exposure levels (6 weeks) by placing a dosimeter inside the incubator
Other: Follow-up of daily infants environmental and clinical parameters — Follow-up of daily infants environmental and clinical parameters: morphological characteristics, drugs, ventilatory support, dietary management, clinical outcomes, incubator data (temperatures…)
Other: Nocturnal polysomnography — Nocturnal polysomnography (at 3 and 6 weeks of life, between 8 pm and 8 am) with recording of sleep (electroencephalography, electrooculography),
Diagnostic Test: cerebral hemodynamics — cerebral hemodynamics (near infrared spectroscopy)
Diagnostic Test: activity of the autonomic nervous system — activity of the autonomic nervous system (electrocardiography, analysis of heart rate variability)

SUMMARY:
The massive use of highly technological devices in Neonatal Intensive Care Units may expose preterm neonates to electromagnetic fields, especially radiofrequencies, at low doses but continuously and chronically. Strikingly, the effect of long-term exposure to radiofrequencies on the neurophysiological development of preterm neonates has never been studied so far. The only studies on the impact of chronic exposure to radiofrequencies have been conducted in animals or adult humans, whereas preterm infants may be particularly vulnerable due to increased penetration of radiofrequency waves into the brain during a crucial period of neurodevelopment. The present project will aim at 1) quantifying individual levels of chronic exposure (during 6 weeks) to which preterm neonates are subjected during their stay in the Neonatal Intensive Care Unit, 2) following the evolution of the thermal environment and of the clinical parameters of the neonates after birth, 3) identifying potential alterations of neurophysiological activity (sleep, cerebral hemodynamics, autonomic nervous activity) which will be correlated to actual levels of chronic RF-EMF (radiofrequency electromagnetic fields) exposure.

DETAILED DESCRIPTION:
Preterm infants are potentially exposed to chronic, low levels of electromagnetic fields, especially radiofrequencies, while hospitalized in neonatal intensive care units. Moreover, they may be particularly vulnerable due to increased penetration of radiofrequency waves into the brain during a crucial period of neurodevelopment. This study will aim at evaluating the influence of radiofrequency electromagnetic fields exposure on the neurophysiological development in preterm neonates.

The first part of this study will be devoted to the measurement of environmental electromagnetic fields in order to map their distribution in the paediatric department. From birth and during 6 weeks, the investigators will perform, for each child, a continuous measurement of radiofrequencies at the incubator level. Infants' clinical data (medical history, nutrition, morphology...) and the evolution of the thermal environment in incubators (air and body temperatures) will also be continually monitored. At 3 and 6 weeks of life, the investigators will investigate sleep (EEG, EOG), cerebral hemodynamics (near-infrared spectroscopy), autonomic nervous system activity (ECG, heart rate variability) and various cardiorespiratory parameters (SpO2, apnoea, bradycardia) thanks to a night-time polysomnography.

The impact of radiofrequency electromagnetic fields will be evaluated by analyses of the relationship between exposure levels and the various parameters extracted from the neurophysiological investigation phase.

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates born at 26 to 34 weeks of gestational age
* signed written informed consent form

Exclusion Criteria:

* infants infected
* infants suffering from neurological disorders
* serious heart, respiratory, digestive or metabolic diseases
* infants born from mothers aged less than 18 years old or deprived of their parental rights
* non covered by national health insurance

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
total sleep time in hours | from birth to 6 weeks of life
  Sleep Structure will be determined by measuring total sleep time, absolute and relative durations of sleep states and sleep state change frequency.
absolute durations of sleep states in hours | from birth to 6 weeks of life
  Sleep Structure will be determined by measuring total sleep time, absolute and relative durations of sleep states and sleep state change frequency.
relative durations of sleep states in hours | from birth to 6 weeks of life
  Sleep Structure will be determined by measuring total sleep time, absolute and relative durations of sleep states and sleep state change frequency.
sleep state change frequency | from birth to 6 weeks of life
  Sleep Structure will be determined by measuring total sleep time, absolute and relative durations of sleep states and sleep state change frequency.

SECONDARY OUTCOMES:
Cerebral hemodynamics | from birth to 6 weeks of life
  Cerebral hemodynamics will be determined by measuring regional cerebral oxygen saturation
Autonomic nervous system activity | from birth to 6 weeks of life
  Autonomic nervous system activity will be determined by measuring means of a heart rate variability
apnea frequency | from birth to 6 weeks of life
  cardiorespiratory parameters (apnea, bradycardia, desaturation) will be determined
bradycardia frequency | from birth to 6 weeks of life
  cardiorespiratory parameters (apnea, bradycardia, desaturation) will be determined
desaturation frequency | from birth to 6 weeks of life
  cardiorespiratory parameters (apnea, bradycardia, desaturation) will be determined
Evolution of the anthropomorphic characteristics of the subjects | from birth to 6 weeks of life
  anthropomorphic characteristics of the subjects are height and weight. Weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tourneux, Pr, Principal Investigator — CHU Amiens; François Moreau, MD, Principal Investigator — CHU Amiens; Lucie Aimée Razafimanantsoa, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No